CLINICAL TRIAL: NCT06035705
Title: Patient Acuity Measures as Part of Daily Managment: a Mixed-methods Study Within Somatic In-patient Care
Brief Title: Patient Acuity in Somatic In-patient Care
Status: Recruiting | Type: Observational
Sponsor: Region Gävleborg (Other)
Collaborators: University of Gavle (Other)
Responsible Party: Sponsor
Other Study IDs: 280936
Record Dates: First submitted 2023-07-07; First posted 2023-09-13 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Work Related Stress
Keywords: nurse staffing; acuity; workload; daily management; job satisfaction
MeSH Terms: conditions — Occupational Stress

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Patient acuity tool — A tool for measuring patient acuity as a part of daily management will be implemented in four somatic in-patient care units.

SUMMARY:
This study addresses nursing acuity measures within somatic in-patient care. Quantitative and qualitative analyses will be used in order to examine staffing levels and nurses' perception of work environment, before, during and after the implementation of a patient acuity tool as a part of daily management.

DETAILED DESCRIPTION:
Nurses' work environment is associated with both quality of care and organizational outcomes. There is a clear relationship between nurse staffing and both patient outcomes and nurses' perception of work environment. The severity of patients' illness is not sufficient for making nurse assignment decisions. One benchmark of staffing is valid measurement of patient acuity (patients' nursing care needs). Patient acuity measures offer a potential for real-time matching of patient demand for nursing care. It is defined as a measure of the severity of illness and the nursing care needs, complexity, and workload required to provide care to a patient or group of patients.

There is a limited amount of research that examine the process of making direct nurse staffing deicions in relation to patient acuity. By examining staffing levels and nurses' perception of work environment in relation to measured patient acuity, we hope to contribute to this field.

The overall aim of this research project is to examine patient-acuity measures as a part of daily management, as being introduced to five wards within the somatic in-patient care in Gävleborg County, Sweden in autumn 2023. The studies will focus on staffing levels in relation to the patient acuity scores and on nurses' perception of work environment, both before, during and after the start of the new work procedures, but also on a weekly basis, related to the acuity scores of the actual work shift.

Data will be collected before, 6 months, and12 months after the implementation of patient acuity measures, using a web-based survey that reaches all the nursing staff at the wards. Data will be analysed with descriptive and inference statistics to explore if the novel work process has brought differences of different asopects related to the nurses' work environment such as their well-being and perception of stress. As a reference, the same procedures will be carried out at two wards that haven't implemented patient acuity measures.

Patient-acuity measures will be collected two times a day (morning and evening shifts) from each of the five wards. Once a week, all nurses working at a particular shift will be asked to make a short estimation (through a paper-based form) of their perception of the work environment during that particular shift. These estimations with single item-measures will be compared with the patient acuity and actual staffing during the shift. An index will be used to compare staffing and patient acuity in the five wards.

Furthermore, semi-structured interviews with four nurses' and the manager from each ward will be conducted with the same time intervals as the web-based surveys. Results will be analysed with content analysis.

ELIGIBILITY:
Inclusion Criteria:

* All nurses employed by the medical wards
* First-line managers at each ward

Exclusion Criteria:

* Travelling nurses
* Nurses with <1 months employment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Nurses here refer to both trained nurses and assistant nurses.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-09-30 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Workplace environment | Baseline measure during November 2021
  Questions on work environment will be asked through a survey. The survey contains questions from the following questionnaires: Conditions of Work Effectiveness Questionnaire (CWEQ-II), Copenhagen Psychosocial Questionnaire (COPSOQ), Thriving Scale and Staff Satisfaction with Care (SSC).
  CWEQ-II: Values between 1-5. Higher scores mean a better outcome in factors on perceived access to opportunity, support, information and resources in an individual's work setting.
  COPSOQ: Values between 1-5. Higher scores mean a better outcome in factors on stress and emotional demands, but a worse outcome in factors on workplace community and involvement, with one item reversed.
  SSC: Values between 1-7. Higher scores mean a better outcome.
  Thriving Scale: Values between 1-7. Higher scores means a better outcome, with one item reversed.
Workplace environment | Measures will be made approximately in June 2024.
  Questions on work environment will be asked through a survey. The survey contains questions from the following questionnaires: Conditions of Work Effectiveness Questionnaire (CWEQ-II), Copenhagen Psychosocial Questionnaire (COPSOQ), Thriving Scale and Staff Satisfaction with Care (SSC).
  CWEQ-II: Values between 1-5. Higher scores mean a better outcome in factors on perceived access to opportunity, support, information and resources in an individual's work setting.
  COPSOQ: Values between 1-5. Higher scores mean a better outcome in factors on stress and emotional demands, but a worse outcome in factors on workplace community and involvement, with one item reversed.
  SSC: Values between 1-7. Higher scores mean a better outcome.
  Thriving Scale: Values between 1-7. Higher scores means a better outcome, with one item reversed.
Workplace environment | Measures will be made approximately during December 2024.
  Questions on work environment will be asked through a survey. The survey contains questions from the following questionnaires: Conditions of Work Effectiveness Questionnaire (CWEQ-II), Copenhagen Psychosocial Questionnaire (COPSOQ), Thriving Scale and Staff Satisfaction with Care (SSC).
  CWEQ-II: Values between 1-5. Higher scores mean a better outcome in factors on perceived access to opportunity, support, information and resources in an individual's work setting.
  COPSOQ: Values between 1-5. Higher scores mean a better outcome in factors on stress and emotional demands, but a worse outcome in factors on workplace community and involvement, with one item reversed.
  SSC: Values between 1-7. Higher scores mean a better outcome.
  Thriving Scale: Values between 1-7. Higher scores means a better outcome, with one item reversed.

SECONDARY OUTCOMES:
Point estimations on workload and patient acuity | Weekly measures from November 2023 to December 2024
  Short protocol involving questions about patient acuity measures in relation to the workshift. The point estimation includes questions about workload, patient safety, staffing, patient acuity. Values between 1 and 10 where higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Region Gävleborg, Gävle, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Brennan CW, Daly BJ. Methodological challenges of validating a clinical decision-making tool in the practice environment. West J Nurs Res. 2015 Apr;37(4):536-45. doi: 10.1177/0193945914539738. Epub 2014 Jun 18. PMID 24948588
- [Result] Engstrom M, Martensson G, Palsson Y, Stromberg A. What relationships can be found between nurses' working life and turnover? A mixed-methods approach. J Nurs Manag. 2022 Jan;30(1):288-297. doi: 10.1111/jonm.13494. Epub 2021 Nov 7. PMID 34643314
- [Result] Debergh DP, Myny D, Van Herzeele I, Van Maele G, Reis Miranda D, Colardyn F. Measuring the nursing workload per shift in the ICU. Intensive Care Med. 2012 Sep;38(9):1438-44. doi: 10.1007/s00134-012-2648-3. Epub 2012 Aug 9. PMID 22875336
- [Result] Eastman D, Kernan K. A New Patient Acuity Tool to Support Equitable Patient Assignments in a Progressive Care Unit. Crit Care Nurs Q. 2022 Jan-Mar 01;45(1):54-61. doi: 10.1097/CNQ.0000000000000388. PMID 34818298